CLINICAL TRIAL: NCT03993613
Title: Efficacy and Safety of Human Apotransferrin in Patients With β-thalassemia Intermedia
Brief Title: Apotransferrin in Patients With β-thalassemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: no availability of IMP for this study
Sponsor: Prothya Biosolutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MD2014.01
Record Dates: First submitted 2019-05-29; First posted 2019-06-20 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: β-thalassemia Intermedia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- human apotransferrin (Experimental): Patients will receive an intravenous dose of human apotransferrin every two weeks for 14-18 weeks.
  Interventions: Biological: human apotransferrin

INTERVENTIONS:
Biological: human apotransferrin — Intravenous infusions

SUMMARY:
The aim of the trial is to study the effect of apotransferrin administration in patients suffering from β-thalassemia intermedia in order to restore the erythropoiesis as reflected by enhanced haemoglobin levels or reduced transfusion dependency.

ELIGIBILITY:
Inclusion Criteria:

* Non-transfusion dependent β-thalassemia intermedia, defined as patients with microcytic anaemia in combination with an elevated HbA2 (>2.5%) and a haemoglobin of <6.2 mmol/L, or transfusion dependent β-thalassemia treated with a regular transfusion schedule.
* Age above≥ 17 years.
* Adequate renal and hepatic function tests
* WHO performance 0, 1 or 2.
* Signed informed consent.

Exclusion Criteria:

* Known with allergic reactions against human plasma or plasma products.
* Concurrent severe and/or uncontrolled medical condition (e.g. uncontrolled diabetes, infection, hypertension, pulmonary disease).
* Cardiac dysfunction as defined by: myocardial infarction within the last 6 months of study entry, unstable angina, or unstable cardiac arrhythmias.
* Pregnant or lactating females.
* Known with IgA deficiency with anti-IgA antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Erythropoiesis | 17 weeks
  Change of haemoglobin level and/or or change of number of RBC units transfused/week

SECONDARY OUTCOMES:
Change from baseline in serum iron | 17 weeks
Change from baseline in change plasma levels of advanced glycation end products | 17 weeks
Change in spleen size | at baseline and at 16 weeks
Change from baseline in reticulocyte count | 17 weeks
Change from baseline in erythropoietin levels | 17 weeks
Ctrough | predose and postdose 5 minutes, 2 hours and 1, 4, 7, 14 days
  Ctrough calculated from serum transferrin levels
Cmin | predose and postdose 5 minutes, 2 hours and 1, 4, 7, 14 days
  Cmin calculated from serum transferrin levels
tmax | predose and postdose 5 minutes, 2 hours and 1, 4, 7, 14 days
  tmax calculated from serum transferrin levels
Cmax | predose and postdose 5 minutes, 2 hours and 1, 4, 7, 14 days
  Cmax calculated from serum transferrin levels
AUCτ | predose and postdose 5 minutes, 2 hours and 1, 4, 7, 14 days
  AUCτ calculated from serum transferrin levels
Ctrough | predose
  Ctrough calculated from serum transferrin levels
Adverse events | 17 weeks
  Number of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Bart Biemond, MD, PhD, Principal Investigator — Academic Medical Centre
Locations (1):
- Academic Medical Centre, Amsterdam-Zuidoost, North Holland, Netherlands